CLINICAL TRIAL: NCT07071402
Title: A Single-center, Single-arm, Open Study on the Treatment of Early Small Breast Cancer With Ultrasound-guided Vacuum-assisted Excision Combined With Surgery
Brief Title: A Study on the Treatment of Early Small Breast Cancer With Ultrasound-guided Vacuum-assisted Excision Combined With Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY-20252227-F-1
Record Dates: First submitted 2025-06-29; First posted 2025-07-17 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer (Early Breast Cancer)
Keywords: vacuum-assisted excision
MeSH Terms: conditions — Breast Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Ultrasound-guided VAE combined with surgery for the treatment of early small breast cancer (Experimental): Single early breast cancer subjects with Tis (carcinoma in situ) or T1 (maximum tumor diameter ≤2cm) and negative axillary lymph nodes on imaging, after being fully informed and signing the informed consent form, and passing the screening, enter the trial period. After the subjects are confirmed to be enrolled, VAE is performed first. Patients with a clear diagnosis of breast cancer receive traditional radical mastectomy for breast cancer: Breast-conserving surgery or total mastectomy, and sentinel lymph node biopsy or dissection in the axilla. The complete resection of the lesion is evaluated based on the postoperative pathology, and follow-up is conducted.
  Interventions: Procedure: Ultrasound-guided vacuum-assisted excision combined with surgical treatment

INTERVENTIONS:
Procedure: Ultrasound-guided vacuum-assisted excision combined with surgical treatment — Patients undergoing VAE surgery （EnCor® vacuum-assisted minimally invasive rotary system）are placed in an appropriate position, undergo routine disinfection and blanching, and the tumor location is located by ultrasound. After local anesthesia, a vacuum-assisted rotary cutting needle is percutaneous punctured beneath the tumor. Under ultrasound guidance, the tumor tissue is gradually resected until the ultrasound shows complete tumor resection. The resected tissue is sent for pathological examination. After the patient is confirmed to have breast cancer through VAE resection biopsy, depending on the patient's specific condition, they are hospitalized for radical mastectomy. The surgical methods can be breast-conserving surgery or mastectomy. At the same time, sentinel lymph node biopsy is performed, and the resected tissue is sent for pathological examination. The surgical process follows the surgical treatment norms for breast cancer.

SUMMARY:
The aim of this clinical trial is to assess the feasibility and safety of ultrasound-guided vacuum-assisted excision (VAE) in the treatment of early breast cancer with Tis (carcinoma in situ) or T1 (maximum tumor diameter ≤2cm) and negative axillary lymph nodes on imaging. The main question it aims to answer is:

* After VAE, when undergoing routine breast cancer surgery again, what is the complete resection rate of the lesion in the surgically removed tissue (pathologically confirmed), that is, the false negative rate of VAE?
* Which type of breast cancer lesion has the highest complete resection rate?
* Is it clear whether VAE can be applied in the treatment of early breast cancer with Tis or T1 and negative axillary lymph nodes on imaging?
* Do patients with benign breast nodules who undergo VAE or are recommended for Vacuum-assisted breast biopsy (VABB) due to limited puncture and are diagnosed with breast cancer need to undergo surgery again?
* The incidence of complications of VAE.

Participants will:

* Single early breast cancer subjects with Tis or T1 and negative axillary lymph nodes on imaging, after being fully informed and signing the informed consent form, enter the trial period after screening and being qualified.
* After the subjects are confirmed to be enrolled, VAE biopsy resection is performed first.
* Patients clearly diagnosed with breast cancer receive traditional radical mastectomy for breast cancer: Breast-conserving surgery or total mastectomy, sentinel lymph node biopsy or dissection in the axilla, assessment of whether the lesion has been completely removed based on postoperative pathology, and follow-up is conducted.

DETAILED DESCRIPTION:
This is a single-arm and single-center clinical study. The specific implementation steps of the study are as follows:

1. Patient recruitment and screening Recruit eligible patients through channels such as the breast surgery outpatient department of the hospital. Conduct a preliminary assessment of potential patients, including medical history inquiry, physical examination, and imaging examinations (breast ultrasound, mammography, etc.), to determine whether they meet the inclusion criteria. Adopt the Common Decision Questionnaire (SDM-Q-9).

   Evaluate the patients and select those with better compliance and a standardized total score of the scale ≥80. Introduce in detail the research purpose, methods, risks and benefits, etc. to the patients who meet the inclusion criteria and the assessment, and obtain the written informed consent forms of the patients.
2. VAE surgery Ultrasound-guided vacuum-assisted resection: Place the patient in an appropriate position, and use a routine disinfection towel. Locate the tumor location by ultrasound. After local anesthesia, percutaneously puncture a vacuum-assisted rotary cutting needle beneath the tumor. Under ultrasound guidance, gradually remove the tumor tissue until the ultrasound shows that the tumor is completely resected. Send the resected tissue for pathological examination.
3. Follow-up surgery After the patient is confirmed to have breast cancer through VAE resection biopsy, according to the specific condition of the patient, perform radical mastectomy for breast cancer in the hospital. The surgical methods can be breast-conserving surgery or mastectomy. At the same time, perform sentinel lymph node biopsy, and send the resected tissue for pathological examination. The surgical process follows the procedures for breast cancer surgical treatment norms.
4. Postoperative assessment Pathological assessment: Conduct a detailed pathological examination on the specimens removed by vacuum-assisted resection and subsequent surgical resection, including tumor size, histological grade, molecular typing, resection margin conditions, and tumor residue conditions, etc.

   Complication assessment: Observe whether complications such as bleeding, infection, breast tissue injury, poor incision healing, and lymphatic leakage occur in patients during vacuum-assisted resection and subsequent surgeries. Record the occurrence time, severity, and treatment measures of complications. Evaluation of surgical satisfaction, treatment satisfaction and quality of life satisfaction: After the operation, give chemotherapy, targeted therapy or endocrine therapy according to the diagnosis and treatment routine. The treatment plan follows the recommendations of guidelines such as NCCN. If local radiotherapy is required, carry it out according to the clinical routine. At 1 week, 1 month, 3 months and 6 months after the operation at time points such as months, evaluate the surgical satisfaction, treatment satisfaction and quality of life satisfaction of the patients.
5. Establish a database for follow-up Utilize the existing breast cancer database of the department to establish individual information data for patients, recording their general information, diagnosis and treatment processes, and other data.

ELIGIBILITY:
Inclusion criteria：

Subjects must meet all of the following inclusion criteria to be enrolled in this trial:

* Age: 18 - 70 years old;
* Female patients;
* Patients diagnosed with suspected breast cancer through imaging (such as breast ultrasound, mammography, etc.) with BI - RADS Category 4C and Category 5;
* Clinical stage T1: Mass ≤2cm;
* No previous treatment related to breast cancer;
* Be willing to undergo ultrasound - guided vacuum - assisted resection, biopsy and surgical treatment; 7) The subjects voluntarily join this study and sign the informed consent form.

Exclusion criteria：

Those with any of the following circumstances will not be selected as subjects:

* Imaging suggests that the lesion is greater than 2cm;
* Suspected positive axillary lymph nodes in imaging (Bedi 4, Bedi 5, Bedi 6);
* The tumor invades the nipples, areolas and subcutaneous tissues;
* Breast cancer during pregnancy;
* Abnormal functions of vital organs such as the heart, lungs, liver and kidneys, and poorly controlled diabetes, etc., cannot tolerate surgery;
* Any other circumstances in which the researcher deems the patient unsuitable to participate in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
The complete resection rate of the lesion in the surgically resected tissue after vacuum-assisted excision under ultrasound guidance | Two weeks after the operation
  The proportion of patients whose tumor tissues are completely resected by VAE confirmed through postoperative pathological examination, that is, the false negative rate of VAE

SECONDARY OUTCOMES:
Incidence of surgery-related complications | During the operation, 3 days after the operation, 2 weeks after the operation, 1 month after the operation
  The occurrence of complications such as bleeding, infection, breast tissue injury, poor incision healing and lymphatic leakage during VAE and subsequent surgical procedures
The local recurrence rate of the breast and axilla | Two years after the operation
  The patients are followed up to evaluate whether there is recurrence of breast and axillary lesions
Patient satisfaction | Three months after the operation
  The BREAST Q2 questionnaire is used for the investigation

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided